CLINICAL TRIAL: NCT03579095
Title: Investigating the Acute and Chronic Effects of an American Ginseng Root Extract on Cognition and Mood.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Naturex (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Chair of Neuroscience, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RDG-004
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Cognitive Change; Effects of Ginseng on Cognitive Function
MeSH Terms: interventions — Cereboost; Asian ginseng

STUDY DESIGN:
Intervention Model Description: Between and within groups model
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- American ginseng (Experimental): 200mg Cereboost and Maltodextrin
  Interventions: Dietary Supplement: Cereboost
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cereboost — 200mg Cereboost and Maltodextrin capsules
  Other Names: American ginseng
  Arms: American ginseng
Dietary Supplement: Placebo — 200mg Maltodextrin capsules
  Arms: Placebo

SUMMARY:
Ginseng refers to the extract of any slow growing perennial plant with a fleshy root, deriving from the Panax genus of the Araliaceae family. Ginseng root has been used as an intervention for the treatment of diabetes (Sotaniemi, Haapakoski & Rautio, 1995), boosting cognitive function (Scholey et al., 2010) and improving mental health (Ellis & Reddy, 2002). The most commonly used ginseng is Panax ginseng (Asia) and Panax quinquefolius (America). Ginsensosides are considered the core phytochemical compounds that contribute to the alleged beneficial effects of ginseng. In particular, ginsenosides Rb1 and Rg1 have been isolated and investigated for effects on cognitive function (Shin et al., 2016).

Scholey et al. (2010) was one of the first studies to provide support for a beneficial cognitive effect from American ginseng (Cereboost™), with better performance on working memory in healthy young adults. Improvements were most profound for a single dose of 200 mg on working memory tasks, specifically immediate word recall and numeric working memory speed. Cereboost also increased self-rated calmness compared to placebo, suggesting ginseng can enhance aspects of mood. Similarly, Ossoukhova et al. (2015) compared a single 200mg dose to placebo to investigate whether beneficial cognitive effects extend to a middle-aged cohort. Here, Cereboost significantly improved performance on the Cognitive Drug Research (CDR) working memory factor, specifically improving spatial working memory at three hours post dose.

Further study is required to evaluate ginseng specific effects with a standardized extract of P. quinquefolius, such as Cereboost™ on healthy participants. Significant results will have implications for investigating the neurocognitive effects in other populations, such as those with cognitive and memory problems.

DETAILED DESCRIPTION:
The study comprises of a familiarisation visit and then two test days. The test days are separated by a 2 week interval during which time participants will be asked to consume a daily capsule for 14 days which will contain either an American ginseng root extract (200 mg Cereboost and Maltodextrin) or an identical placebo that does not contain any of the active ingredient. Participants will be asked to restrict their intake of certain foods for 48 hours before test days and intake of alcohol and caffeinated drinks for 24 hours prior. All participants will be required to fast overnight prior to each of the study days. Participants may withdraw at any time without giving any reason. In addition, a participant will be withdrawn from the study if they request discontinuation, exhibit a serious adverse event to any component of the test product, the participant significantly violates the exclusion or inclusion criteria, an illness emerges and/or opinion is that withdrawal is appropriate.

An outline of each session is as follows:

1. Familiarisation/practice visit: Volunteers will attend the Nutritional Psychology unit at the University of Reading, where they will receive a detailed explanation on the study and will be asked to sign the informed consent form. Once consent has been given the inclusion/exclusion criteria will be checked and measures of age, height and weight will be taken. Participants will then be asked to fill out a food frequency questionnaire before completing training on the cognitive test battery. Participants will be given two food diaries, with each diary completed in the 48 hours before each test day to check habitual diet and ensure they followed low flavonoid protocol. Finally the PANAS - X will be administered to gain a measure of trait mood
2. Test visits: On arrival of their first test day, participants will be randomly assigned to treatment (200 mg Cereboost™) or placebo condition. Each study day will begin at 9am with breakfast before completion of the computerized test battery to establish baseline performance. Participants will then take their allocated intervention and will be tested on the cognitive and mood battery at 2, 4 and 6 hours after consumption. A standard light lunch will be provided between the 2hr and 4 hr test points. On test visit 2, participants will have completed a 14 day course of their intervention and will be tested at the same time points at test visit 1, again receiving the intervention directly after the baseline test battery. Finally the PANAS - X will be administered again to gain a measure of trait mood following the 2 week intervention.

The computerized cognitive battery will include tests which are known to be sensitive to nutritional manipulations (Lamport, 2012) and will last no more than 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* healthy, between 18-30

Exclusion Criteria:

* Smoke
* Use medications that may affect the outcome
* Have any allergic reactions to ingredients in the capsules
* Have a BMI greater than or equal to 30
* Are vegetarian
* Taking any dietary supplements which they are unwilling to stop for the duration of the study
* Drink more than 2 alcoholic beverages per day on an average week
* Have participated in any other cognitive trials within the last month.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Rapid Visual Information Processing task | 14 Days
  This task will assess attention processes. In this task a series of digits are presented one at a time on the screen, in quick succession at a rate of 100/min. The participant must examine the continuous series for a sequence of three consecutive even or three consecutive odd digits. The participant must respond once they have detected a sequence string by pressing the space bar as quickly as possible. Up to 8 correct target strings will be presented in each minute, and the task will last approximately 6 minutes. The task will be scored for accuracy.

SECONDARY OUTCOMES:
Immediate word recall | 14 Days
  Using the methodology outlined in Scholey et al., (2010), participants will be presented with a sequential list of 15 words, at a rate of 1 word per second. The participant will then have 60s to type as many of these words as possible, with the resulting score recorded as a percentage of accuracy.
Corsi blocks task | 14 Days
  This task examines visuospatial memory. Nine identical squares are fixed in a random arrangement on a screen. Participants observe spatial sequences of between two and nine blocks. Four versions of each sequence length presented during the task. The task is to reproduce the sequence, immediately after each presentation by pressing the relevant squares on the screen. The dependent variable is the number of blocks pointed out in the correct order. A novel sequence will be presented on each occasion, the order of which will be counterbalanced across participants.
Modified Attention Network Task | 14 Days
  This task examines execution function, attention and inhibition. In this task, participants have to respond to a centrally presented arrow, pointing to the left or the right by pressing the corresponding key on the keyboard. The central arrow is flanked by arrows that point in the same (congruent) or opposite (incongruent) direction. In order to perform the task effectively, participants have to ignore the flanking arrows. Previous studies have found that participants show larger latencies and more errors on incongruent trials when compared with congruent trials due to the conflicting interference of the incongruently facing arrows. The response latencies to congruent trials reflect processing speed, while the amount of interference during incongruent trials indicates susceptibility to interference.
Task Switch Task | 14 Days
  This task measures executive function and attention. Participants view a circle with 8 equally spaced radii 2 of which form a bold bisecting line. Numbers are chosen randomly from a set of 1-4 & 6-9 and displayed sequentially in a clockwise direction. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. General measures of accuracy and response time along with specific measures of switching cost for the first trial after each task change are acquired.
Delayed word recall | 14 Days
  Approximately 35 minutes after the immediate word recall task, participants will be allowed 60seconds to write down as many items they can remember from the immediate word recall test.
Mood | 14 Days
  The Positive and Negative Affect Scale (PANAS - N) will be used to examine mood states at the start and end of the cognitive task battery. It is regarded as a reliable measure for non-clinical populations (Crawford et al, 2004). Participants are asked to rate the extent to which they experienced each out of 20 emotions on a 5-point Likert scale ranging from "very slightly" to "very much". Half of the presented emotion words concern negative affect (distressed, upset, guilty, ashamed, hostile, irritable, nervous, jittery, scared, afraid), the other half positive affect (interested, alert, attentive, excited, enthusiastic, inspired, proud, determined, strong, active). Additionally, the PANAS - X will be used to measure trait mood.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Psychology and Clinical Languages, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sotaniemi EA, Haapakoski E, Rautio A. Ginseng therapy in non-insulin-dependent diabetic patients. Diabetes Care. 1995 Oct;18(10):1373-5. doi: 10.2337/diacare.18.10.1373. PMID 8721940
- [Background] Scholey A, Ossoukhova A, Owen L, Ibarra A, Pipingas A, He K, Roller M, Stough C. Effects of American ginseng (Panax quinquefolius) on neurocognitive function: an acute, randomised, double-blind, placebo-controlled, crossover study. Psychopharmacology (Berl). 2010 Oct;212(3):345-56. doi: 10.1007/s00213-010-1964-y. Epub 2010 Jul 31. PMID 20676609
- [Background] Ellis JM, Reddy P. Effects of Panax ginseng on quality of life. Ann Pharmacother. 2002 Mar;36(3):375-9. doi: 10.1345/aph.1A245. PMID 11895046
- [Background] Shin K, Guo H, Cha Y, Ban YH, Seo da W, Choi Y, Kim TS, Lee SP, Kim JC, Choi EK, Yon JM, Kim YB. Cereboost, an American ginseng extract, improves cognitive function via up-regulation of choline acetyltransferase expression and neuroprotection. Regul Toxicol Pharmacol. 2016 Jul;78:53-8. doi: 10.1016/j.yrtph.2016.04.006. Epub 2016 Apr 22. PMID 27112419
- [Background] Ossoukhova A, Owen L, Savage K, Meyer M, Ibarra A, Roller M, Pipingas A, Wesnes K, Scholey A. Improved working memory performance following administration of a single dose of American ginseng (Panax quinquefolius L.) to healthy middle-age adults. Hum Psychopharmacol. 2015 Mar;30(2):108-22. doi: 10.1002/hup.2463. PMID 25778987
- [Derived] Bell L, Whyte A, Duysburgh C, Marzorati M, Van den Abbeele P, Le Cozannet R, Fanca-Berthon P, Fromentin E, Williams C. A randomized, placebo-controlled trial investigating the acute and chronic benefits of American Ginseng (Cereboost(R)) on mood and cognition in healthy young adults, including in vitro investigation of gut microbiota changes as a possible mechanism of action. Eur J Nutr. 2022 Feb;61(1):413-428. doi: 10.1007/s00394-021-02654-5. Epub 2021 Aug 15. PMID 34396468